CLINICAL TRIAL: NCT04419298
Title: Evaluation for Acute and Chronic Features of Cardiac Injury by CMR in Acute CO Poisoned Patients With Elevated Troponin I (TnI)
Brief Title: Cardiac Magnetic Resonance Image (CMR) in Acute Carbon Monoxide (CO) Poisoning
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: CMR-CO
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Carbon Monoxide Poisoning; Myocardial Injury; Image, Body
MeSH Terms: conditions — Carbon Monoxide Poisoning | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute CO poisoning with myocardial injury: A diagnosis of CO poisoning was made according to medical history and carboxyhaemoglobin >5% (>10% in smokers).
  Myocardial injury was defined as elevated high-sensitivity TnI level above the upper limit (> 0.046 ng/mL) when measured in the emergency department (ED) or repeatedly within 24 hours after ED arrival.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — 1. Cardiac MRI be taken to acute CO poisoned patients with elevated TnI [during acute (within 7 days after CO exposure) and chronic phase (at 4-5 months after CO exposure)]
  2. TTE be taken to acute CO poisoned patients with elevated TnI [At the ED and during admission (within 7 days after CO exposure)]
  Other Names: Transthoracic echocardiography (TTE)

SUMMARY:
Previous report showed that 37% of patients with moderate to severe carbon monoxide (CO) poisoning experienced a myocardial injury, defined as elevated cardiac enzyme [creatine kinase, CK-MB, and cardiac troponin I (TnI)] or ischemic electrocardiogram (ECG) change. In other study, 24% of the patients with the myocardial injury after CO poisoning died during a median follow-up of 7.6 years. The myocardial injury was the major predictor of mortality. In addition, in the Taiwanese nationwide population-based cohort study, CO poisoning itself reported as a higher risk of a major adverse cardiovascular event.

According to the previous study of investigators, among CO poisoned patients with myocardial injury, 74.4% of patients experienced CO-induced cardiomyopathy. All CO-induced cardiomyopathy recovered to normal status. In this situation, there is no definite approved reason why more cardiovascular events are occurred in CO poisoned patients with myocardial injury during long term follow-up period despite normalization of CO-induced elevated TnI and cardiac dysfunction.

Two image cases related to cardiac magnetic resonance imaging (CMR) in acute CO poisoning previously reported. One image case reported that patient had mildly depressed left ventricular (LV) systolic function with hypokinesis of the anterior wall and regional akinesis of the inferior wall on the transthoracic echocardiography performed during hospitalization and late gadolinium-enhancement (LGE) images of CMR demonstrated multiple focal areas of high signal consistent with myocardial necrosis or fibrosis. Another image case reported an image case that in CMR, inferolateral mid-wall myocardial fibrosis, which was defined as LGE, was present despite the setting of a completely normal echocardiogram at 4-month follow-up in CO poisoned patients.

Therefore, the investigators evaluate prevalence (frequency of LGE positive) and patterns (involved LV wall and range of LGE positive) of myocardial fibrosis (LGE positive) in acute CO-poisoned patients during acute (within seven days after CO exposure) and chronic phase (at 4-5 months after CO exposure) and whether LGE positive developed in acute phase have been changed through cardiac MRI performed at chronic phase. The investigators also evaluate LV ejection fraction and global longitudinal strain in transthoracic echocardiography performed at the ED (baseline) and within seven days (follow-up). The investigators also assessed the association between neurocognitive outcomes using the global deterioration scale (at 1, 6, and 12 months after CO exposure) and the presence of LGE positive.

DETAILED DESCRIPTION:
In the US, carbon monoxide (CO) poisoning accounts for 1,300 deaths and 50,000 emergency department visits annually. Previous report showed that 37% of patients with moderate to severe CO poisoning experience a myocardial injury defined as elevated cardiac enzyme [creatine kinase, CK-MB, and cardiac troponin I (TnI)] or ischemic electrocardiogram (ECG) change. In other study, there was a mortality of 24% of patients during a median follow-up of 7.6 years. A mortality among the patients who experienced the myocardial injury was higher than patients without the myocardial injury. The death caused by cardiovascular problems occurred more among patients with a history of the myocardial injury (44% vs. 18%). The myocardial injury was the major predictor of mortality. In addition, in the Taiwanese nationwide population-based cohort study, a history of CO poisoning showed a higher risk of a major adverse cardiovascular event.

The investigators reported that myocardial injury (defined as elevated TnI or change of ischemic ECG) developed in 20% of CO poisoned patients and elevated TnI was normalized within 65.0 hours. According to previous study of the investigators, among CO poisoned patients with myocardial injury, 74.4% of patients experienced CO-induced cardiomyopathy. All CO-induced cardiomyopathy recovered to normal status. In this situation, there is no definite approved reason why more cardiovascular events are occurred in CO poisoned patients with myocardial injury during long term follow-up period despite normalization of CO-induced elevated TnI and cardiac dysfunction.

One case reported an image related to a CO poisoned patient with acute myocardial injury found by cardiac magnetic resonance imaging (CMR) with a normal coronary artery confirmed by coronary angiography. In that case, a patient showed that patient had mildly depressed left ventricular (LV) systolic function with hypokinesis of the anterior wall and regional akinesis of the inferior wall on the transthoracic echocardiography performed during hospitalization and late gadolinium-enhancement (LGE) images of CMR demonstrated multiple focal areas of high signal consistent with myocardial necrosis or fibrosis. Through this case, the investigators thought that CO poisoning might result in acute myocardial necrosis, demonstrating another type of myocardial injury that can be detected by CMR. In addition, Other case reported an image case that in cardiac MRI, inferolateral mid-wall myocardial fibrosis, which was defined as LGE, was present despite the setting of a completely normal echocardiogram at 4-month follow-up in a patient who experienced severe CO poisoning.

Mid-wall myocardial fibrosis has been reported in dilated cardiomyopathy (DCMP) of unclear origin. In a follow-up study of 101 consecutive patients with DCMP, mid-wall fibrosis (presented in 35% of patients) predicted a combined endpoint of all-cause mortality, cardiovascular hospitalization, and sudden cardiac death. Myocardial fibrosis has also been demonstrated in hypertrophic cardiomyopathy. The myocardial fibrosis has been linked to known markers for sudden cardiac death, although the independent prognostic value of CMR has yet to be determined.

Through above results, the investigators thought that the normal LV cardiac function may not reflect that there is no problem with the heart, and it could lead to myocardial fibrosis in the chronic phase. Myocardial damage seen through CMR may be related to the patient's prognosis. Therefore, the investigators evaluate prevalence (frequency of LGE positive) and patterns (involved LV wall and range of LGE positive) of myocardial fibrosis (LGE positive) in acute CO-poisoned patients during acute (within 7 days after CO exposure) and chronic phase (at 4-5 months after CO exposure) and whether LGE positive developed in the acute phase has been changed in cardiac MRI performed at chronic phase. The investigators also evaluate LV ejection fraction and global longitudinal strain in transthoracic echocardiography performed at the ED (baseline) and within seven days (follow-up). The investigators also assessed the association between neurocognitive outcomes using the global deterioration scale (at 1, 6, and 12 months after CO exposure) and the presence of LGE positive.

ELIGIBILITY:
Inclusion Criteria:

* Acute CO poisoning with myocardial injury, which was defined as elevated TnI (reference range < 0.045 ng/mL), within 24 hours after ED arrival.

Exclusion Criteria:

* Age <19 years
* No elevated TnI within 24 hours after ED arrival
* Cardiac arrest upon ED arrival or before taking a CMR
* Co-ingestion of cardiac toxic drugs
* Transferred patients without admission
* Declined to enrollment in the study
* Impossible CMR due to artificial device
* Calculated creatinine clearance (Ccr) < 30 mL/min
* Previous known history of hypersensitivity of gadolinium
* History of acute coronary syndrome, heart failure, or cardiomyopathy
* Patients who refuse CMR or fail to take a CMR although written informed consent was obtained
* Impossible of interpretation of CMR although CMR was taken

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute CO poisoning with myocardial injury, which was defined as elevated TnI (reference range < 0.045 ng/mL), within 24 hours after ED arrival.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Late gadolinium enhancement (LGE) in CMR | Within 7 days after acute CO poisoning
  Prevalence (percent) of presence of LGE in CMR
LGE involved wall in CMR | Within 7 days after acute CO poisoning
  Injured left ventricular wall according to LGE in CMR

SECONDARY OUTCOMES:
LGE size in CMR | Within 7 days after acute CO poisoning
  Injury size according to LGE in CMR
Change of LGE between first CMR and follow-up CMR | Within 7 days after CO exposure and at 4-5 months after CO exposure
  Change of LGE between first CMR (within 7 days after CO exposure) and follow-up CMR (at 4-5 months after CO exposure)
LV ejection fraction (EF) of TTE performed at the ED | Within 3 hours at the ED
  Baseline LV EF of TTE performed at the ED
LV global longitudinal strain (GLS) of TTE performed at the ED | Within 3 hours at the ED
  Baseline LV GLS of TTE performed at the ED
LV EF of TTE performed during admission | Within 7 days after CO exposure
  Follow-up LV EF of TTE performed during admission
LV GLS of TTE performed during admission | Within 7 days after CO exposure
  Follow-up LV GLS of TTE performed during admission
Change of LV EF between ED TTE and follow-up TTE | Within 3 hours at the ED and within 7 days after CO exposure
  Change of LV EF between baseline TTE and follow-up TTE
Change of LV GLS between ED TTE and follow-up TTE | Within 3 hours at the ED and within 7 days after CO exposure
  Change of LV GLS between baseline TTE and follow-up TTE
Correlation between presence of LGE and poor neurocognitive outcome at 1, 6, and 12 months | GDS (minimum 1 - maximum 7) evaluated at 1, 6, and 12 months after CO exposure
  Correlation between presence of LGE and poor neurocognitive outcome [global deterioration scale (GDS) 4-7] evaluated by GDS at 1, 6, and 12 months after CO exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho DH, Ko SM, Son JW, Park EJ, Cha YS. Myocardial Injury and Fibrosis From Acute Carbon Monoxide Poisoning: A Prospective Observational Study. JACC Cardiovasc Imaging. 2021 Sep;14(9):1758-1770. doi: 10.1016/j.jcmg.2021.02.020. Epub 2021 Apr 14. PMID 33865788